CLINICAL TRIAL: NCT01851954
Title: Pharmacokinetic Study of Clarithromycin in Premature Infants With Safety Evaluation
Brief Title: Pharmacokinetic Study of Clarithromycin in Very Low Birth Weight (VLBW)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: declined enrollment
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Han-Suk Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: clarith_VLBW
Record Dates: First submitted 2013-04-12; First posted 2013-05-13 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Very Low Birth Weight Infant; Ureaplasma/Mycoplasma Positive
MeSH Terms: interventions — Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- clarithromycin (Experimental): Population PK
  Interventions: Drug: Clarithromycin

INTERVENTIONS:
Drug: Clarithromycin — IV clarithromycin infusion

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics of clarithromycin which is used for premature infants with ureaplasma.

ELIGIBILITY:
Inclusion Criteria:

* birthweight < 1500gm or GA < 32 weeks
* transtracheal aspirate/gastric juice ; ureaplasma/mycoplasma(+)

Exclusion Criteria:

* sepsis, hypotension, shock
* major congenital anomaly

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2013-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics | 72 hours after first infusion
  AUC, Cmax

CONTACTS AND LOCATIONS:
Overall Officials: Han-Suk Kim, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Children's Hospital, Seoul, South Korea